CLINICAL TRIAL: NCT00198744
Title: Efficacy of Parent-Child Dieting Plans Incorporating Medifast Meal Replacements for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Medifast, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDI2004-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Eating

INTERVENTIONS:
Behavioral: Medifast FIT! for Kids
Behavioral: standard recommendations for dietary intake in children
Behavioral: both diet plans with and without a parent dieting

SUMMARY:
1. Does a joint parent-child dieting approach, as opposed to an individually-based approach, improve weight loss outcomes?
2. Is a diet which includes Medifast meal replacements as efficacious as a non-supplemented Food Guide Pyramid-based diet (reference diet) in achieving better adherence to the diet, initial weight loss, reduction in % body fat, and weight maintenance?
3. Does regular use of Medifast meal replacements, in conjunction with a Food Guide Pyramid-based diet, result in significantly better compliance, greater dietary satisfaction, dietary quality, and palatability than the reference diet?
4. Do children who have lost weight using Medifast meal replacements, as an adjunct to a Food Guide Pyramid-based diet, achieve health benefits compared to baseline values and are these health benefits greater than those obtained following the reference diet?

DETAILED DESCRIPTION:
Weight Loss Phase: This phase will take place between week 0 and week 26 (6 months). Participants will be randomly assigned to one of two weight loss treatment groups:

1. Medifast meal replacement diet group (3 supplements per day) plus food-based diet
2. Reference diet group (Food Guide Pyramid-based diet)

Participants will be further randomly assigned to one of two parent-child approaches:

1. Dieting child with one dieting parent
2. Dieting child without dieting parent Although it is encouraged to have both parents involved in the child's care, only one parent will be permitted to be dieting as a part of the study along with the child so that we can more cleanly assess the effects of a parent dieting without confounding effects of some families having two parents dieting. Both groups will attend separate biweekly educational lessons during the weight loss phase (same curriculum and teacher). Data collection visits will occur at baseline, week 12, and transition. There are a total of 31 visits for a child participating in this study, and 30.for a parent participating by dieting with their child.

Transition Phase: Transition to a maintenance diet will be individually timed by participant attainment of goal "healthy" weight (BMI≤ 25) or week 26, whichever comes first.

Maintenance Phase: This phase will occur after completion of weight loss or between weeks 27 and 78 (12 months). Groups will attend separate educational lessons (same curriculum and teacher) once every 4 weeks. The Medifast group will reduce supplements to 2 per day with a larger portion of calories from whole foods. The reference diet group will remain on a food-based (no supplements) maintenance diet for the entire 52+ week maintenance period. Data collection visits will occur at weeks 26 and 52.

ELIGIBILITY:
Inclusion Criteria:

1. 80 males and females between 8 and 15 years of age, who are overweight (> 25kg/m2 or BMI > 95th percentile on BMI-for-age growth charts) and desiring weight loss.
2. 40 parents, male or female, with a BMI > 25 kg/m2 and desiring weight loss
3. Not using appetite-affecting medications (e.g. Prozac, Ritalin) unless on established and stable doses
4. Not using weight loss drugs or herbals (phentermine, sibutramine, orlistat, etc…)
5. Willing and able to comply with the protocol requirements
6. Child willing and able to give informed consent/assent
7. Parent or legal guardian willing and able to give informed consent
8. Parents must be willing and able to attend all sessions with the child. (One parent or legal guardian is mandatory, however, both are encouraged to attend.)
9. Have regular source of health care (e.g. pediatrician) and permission of primary care provider

Exclusion Criteria:

1. Uncontrolled or unstable use of medications
2. Chronic uncontrolled health problems (not including obesity, mild dyslipidemia, hypertension <160/95)
3. Bulimia, laxative abuse, substance abuse, alcohol intake > 10 drinks per week, or uncontrolled psychiatric disorder (major depression, bipolar disorder, etc…) as determined at screening
4. Breast-feeding or pregnant at screening (determined by serum pregnancy test when applicable)- If a pregnancy occurs during the protocol treatment will end and the pregnancy will be followed to term.
5. Child/family distress determined by assessment of family situation at screening
6. Food allergies, such as peanuts, to ingredients in Medifast products

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80
Dates: Start 2004-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Weight
BMI

SECONDARY OUTCOMES:
blood changes
body composition
psychometrics

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States